CLINICAL TRIAL: NCT01876043
Title: Efficacy and Safety of Plitidepsin in Patients With Advanced Unresectable or Metastatic, Relapsed/Refractory, Dedifferentiated Liposarcoma (DLPS): an Exploratory Phase II Multicenter Trial
Acronym: APLIPO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: Ministry of Health, France (Other Government); PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IB2011-02
Record Dates: First submitted 2012-10-29; First posted 2013-06-12 (Estimated); Results first posted 2019-11-12 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2020-12

CONDITIONS: Adult Patients With Unresectable Locally Advanced or Metastatic, Relapsed/Refractory Dedifferentiated Liposarcoma
MeSH Terms: conditions — Neoplasm Metastasis; Recurrence; Liposarcoma | interventions — plitidepsin

ARMS (1):
- plitidepsin (Experimental): plitidepsin
  Interventions: Drug: plitidepsin

INTERVENTIONS:
Drug: plitidepsin — Patients received plitidepsin as an i.v. 3-h infusion of 5 mg/m2/day on days 1 and 15 every 4 weeks. Patients discontinued plitidepsin if one of the following occurred: consent withdrawal, unacceptable toxicity, disease progression (RECIST v1.1), intercurrent illness or investigator's decision.
  Single-arm phase II clinical trial based on a two-stage optimal Simon's design with 37 evaluable patients (first stage: 17 patients) used to distinguish a favorable true non-progression rate of 40% from a null rate of 20% (90% power and 10% type I error).
  * Stage 1(17 participants): if <=3 non-progressions at 3 months, the study was stopped early. Otherwise, the second group of 20 participants was recruited.
  * Stage 2 (37 participants): if >= 11 non-progressions, Aplidin was considered promising.

SUMMARY:
Liposarcomas are soft tissue sarcomas most frequent. We distinguish three subtypes on the basis of their histological and cytogenetic characteristics: well-differentiated liposarcoma / dedifferentiated, myxoid liposarcoma and / or round cell liposarcoma and pleomorphic. Dedifferentiated liposarcomas (LDD) represent 20% of liposarcomas and are characterized by well-differentiated component associated with a contingent sarcomatous differentiation and fat-usually high grade. The LDD are most often rétropértionéal seat. Thus, their development is very long asymptomatic. At diagnosis, tumor volume is often very important making surgical removal impossible in a high proportion of cases. Operable tumors have also a risk of local recurrence by about 50% and about 20% metastatic. Chemotherapy is the only treatment of these advanced forms. However, the currently available drugs (adriamycin, ifosfamide) have only very limited effectiveness. Progression-free survival of patients does not exceed 2 months. The LDD is characterized cytogenetically by the constant presence of two amplicons (1p32 and 6q23) respectively targeting genes MAP3K5 and JUN. These two genes encode proteins involved in the signaling pathway Jun N-terminal kinase (JNK). Activation of JNK is involved in the loss of adipose differentiation and tumor aggressiveness of LDD. The plitidepsin is a drug capable of inducing apoptosis of tumor cells carrying a functional activation of the JNK pathway. This drug has such a pro-apoptotic and anti-proliferative in vitro models of LDD. plitidepsin could represent the treatment of choice for patients with advanced LDD. The objective of this study is to evaluate the anti-tumor activity of plitidepsin patients with locally advanced dedifferentiated liposarcomas and / or metastatic.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed and dated written informed consent prior to any study specific procedure.
2. Histologically confirmed DLPS by central review.
3. Metastatic or unresectable locally advanced disease
4. Progressive disease according to RECIST v1.1 criteria diagnosed on the basis of two CT scan obtained at an interval less than 3 months and confirmed by central review
5. At least one prior anthracycline-containing chemotherapy regimen
6. Age ≥ 18 years.
7. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 1.
8. Measurable disease according to RECIST v1.1 outside any previously irradiated field.
9. Adequate hematological, renal, metabolic and hepatic function.

   1. Hemoglobin ≥ 9 g/dl (patients may have received prior red blood cell [RBC] transfusion, if clinically indicated); absolute neutrophil count (ANC) ≥ 1.2 x 109/l, and platelet count ≥ 100 x 109/l.
   2. Alkaline phosphatase (AP), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) 2.5 x upper limit of normality (ULN) (5 in case of extensive skeletal involvement for AP exclusively).
   3. Total bilirubin 1.5 x ULN.
   4. Albumin > 25 g/l.
   5. Calculated creatinine clearance (CrCl) ≥ 40 ml/min (according to cockroft and Gault formula).
   6. Creatine phosphokinase (CPK) ≤ 2.5 x ULN.
10. Troponin I ≤ ULN
11. No prior or concurrent malignant disease in the last 5 years except for adequately treated in situ carcinoma of the cervix, basal or squamous skin cell carcinoma, or in situ transitional bladder cell carcinoma.
12. At least three weeks since last chemotherapy (six weeks in case of nitrosoureas and mitomycin C), immunotherapy or any other pharmacological treatment and/or radiotherapy.
13. Recovery to grade ≤ 1 from any adverse event (AE) derived from previous treatment (excluding alopecia of any grade and non-painful peripheral neuropathy grade ≤ 2) according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE, version 4.0).
14. Left ventricular ejection fraction (LVEF) by echocardiogram (ECHO) or multiple gated acquisition (MUGA) within normal limits.
15. Women of childbearing potential must have a negative serum pregnancy test before study entry. Both women and men must agree to use a medically acceptable method of contraception throughout the treatment period and for six months after discontinuation of treatment. Acceptable methods of contraception include intrauterine device (IUD), oral contraceptive, subdermal implant and double barrier.
16. Patients with a french social security in compliance with the French law relating to biomedical research

Exclusion Criteria:

1. Previous treatment with plitidepsin.
2. More than three prior lines of therapy for advanced disease.
3. Concomitant diseases/conditions:

   1. History or presence of unstable angina, myocardial infarction, congestive heart failure or clinically significant valvular heart disease. Symptomatic arrhythmia or any arrhythmia requiring ongoing treatment, and/or prolonged QT-QTc grade > 1.
   2. Previous mediastinal radiotherapy.
   3. Previous treatment with anthracyclines at cumulative doses in excess of 450 mg/m2 doxorubicin equivalent.
   4. Symptomatic arrhythmia or any arrhythmia requiring ongoing treatment, and/or prolonged QT-QTc grade > 1.
   5. Active uncontrolled infection.
   6. Myopathy or persistent CPK elevations > 2.5 x ULN in two different determinations performed with one week apart.
   7. Any other major illness that, in the Investigator's judgment, will substantially increase the risk associated with the patient's participation in this study.
4. Evidence of progressive or symptomatic central nervous system (CNS) or leptomeningeal metastases.
5. Men or women of childbearing potential who are not using an effective method of contraception as previously described; women who are pregnant or breast feeding.
6. Tumor tissue sample not available for pathological review and/or JNK immunochemistry testing.
7. Participation in a clinical study and / or receipt of an investigational drug during the last 30 days.
8. Previous enrolment in the present study.
9. Patient unable to follow and comply with the study procedures because of any geographical, social or psychological reasons.
10. Known hypersensitivity to any involved study drug or any of its formulation components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Italiano, MD, Study Chair — Institut Bergonié
Locations (6):
- France (6):
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital de la Timone, Marseille
  - Institut Curie, Paris
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Result] Toulmonde M, Le Cesne A, Piperno-Neumann S, Penel N, Chevreau C, Duffaud F, Bellera C, Italiano A. Aplidin in patients with advanced dedifferentiated liposarcomas: a French Sarcoma Group Single-Arm Phase II study. Ann Oncol. 2015 Jul;26(7):1465-70. doi: 10.1093/annonc/mdv195. Epub 2015 Jun 3. PMID 26041763

RESULTS

PARTICIPANT FLOW:
Groups:
- Plitidepsin: Patients received Aplidin® as an i.v. 3-h infusion of 5 mg/m2/day on days 1 and 15 every 4 weeks (q4wk).Patients discontinued Aplidin if one of the following occurred: consent withdrawal, unacceptable toxicity, disease progression (RECIST v1.1), intercurrent illness or investigator's decision.
  Single-arm phase II clinical trial based on a two-stage optimal Simon's design with 37 evaluable patients (first stage: 17 patients) used to distinguish a favorable true non-progression rate of 40% from a null rate of 20% (90% power and 10% type I error).
  * Stage 1(17 participants): if <=3 non-progressions at 3 months, the study was stopped early. Otherwise, the second group of 20 participants was recruited.
  * Stage 2 (37 participants): if >= 11 non-progressions, Aplidin was considered promising.
Period: Overall Study
Arm/Group | Plitidepsin
Started | 24
Interim Analysis Population (Following Simon's 2-stage design (see arm description), 17 patients included in the first stage.) | 17
Completed (Received one complete cycle or two incomplete cycles of treatment (17 patients included in the first stage of Simon's design + 5 additionnal patients included)) | 22
Not Completed | 2
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Plitidepsin
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 10
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63.3 [56.1 to 69.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 12
Region of Enrollment [Number; unit: participants]
  France | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Remaining Alive and Progression Free at 3 Months (i.e. Week 12 ± 1) as Per RECIST1.1 (PFS3).
Description: Progression is defined using New Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of diameters of target lesions (taking as reference the smallest sum on study), or a unequivocal progression of existing non-target lesions, or the appearance of one or more new lesions.
Time Frame: 3 months
Population: 22 patients who completed study i.e who completed one cycle or two incomplete cycles of treatment were analyzed for final efficacy analysis. Out of these 22 patients who completed study, the first 17 patients (first stage of the 2-stage Simon's optimal design ) were analyzed for interim efficacy analysis based on primary endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Plitidepsin
Number analyzed (Participants) | 22
percentage of participants
  Final efficacy analysis | 9.1 [1.1 to 29.2]
  Interim analysis population: number analyzed (Participants) | 17
  Interim analysis population | 5.9 [0.15 to 28.7]

2. Secondary Outcome: Percentage of Patients With Objective Response at Six Months (as Per RECIST v1.1)
Description: Objective response assessed as per New Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) : Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.; Overall Response (OR) = CR + PR.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Plitidepsin
Number analyzed (Participants) | 22
percentage of participants | 0 [0 to 0]

3. Secondary Outcome: Percentage of Patients Remaining Alive and Progression Free at 6 Months as Per RECIST1.1.
Description: as for outcome 1
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Plitidepsin
Number analyzed (Participants) | 22
percentage of participants | 0 [0 to 0]

4. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is defined as the delay between the start date of treatment and the date of progression or death (from any cause), whichever occurs first. Patients alive and progression free were censored at the date of last follow-up, death, or last patient contact. Progression is assessed as per RECIST v1.1.
Time Frame: from start of study treatment to the end of the study (up to 10 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Plitidepsin
Number analyzed (Participants) | 22
months | 1.6 [1.4 to 2.6]

5. Secondary Outcome: 1-year Overall Survival (OS) Rate
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of overall survival
Arm/Group | Plitidepsin
Number analyzed (Participants) | 22
percentage of overall survival | 40.9 [20.9 to 60.1]

6. Secondary Outcome: Treatment Safety (AEs, SAEs and Laboratory Abnormalities) Graded According to the NCI-CTCAE Version 4.0.
Description: Toxicity were graded according to the NCI-CTCAE version 4.0.
Time Frame: through study completion, an average of 1 year
Measure: Number; unit: adverse events
Arm/Group | Plitidepsin
Number analyzed (Participants) | 24
adverse events | 232

7. Secondary Outcome: Number of Participants With a Biomarker Amplification
Description: Genomic status of biomarkers obtained by using array-comparative genomic hybridization.
Time Frame: through study completion, an average of 1 year
Population: 19 patients (out of the 22 patients) for whom translational research have been performed.
Measure: Number; unit: participants
Arm/Group | Plitidepsin
Number analyzed (Participants) | 19
participants | 2

ADVERSE EVENTS:
Arm/Group | Plitidepsin
Serious Adverse Events (participants affected / at risk) | 12/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Plitidepsin (N=24)
ASTHENIA, ANOREXIA, NAUSEA (Metabolism and nutrition disorders) | 1
Diabetic decompensation (Metabolism and nutrition disorders) | 1
CPK increased (Investigations) | 1
Inferior vena cava thrombosis (Vascular disorders) | 1
SUDDEN DEATH (General disorders) | 1
CHEST PAIN / TROPONIN INCREASED (Investigations) | 1
LEFT FOREARM FRACTURE (Injury, poisoning and procedural complications) | 1
WORSENING OF GENERAL STATUS (General disorders) | 1
NAUSEA (Gastrointestinal disorders) | 2
FEVER VOMITING (Gastrointestinal disorders) | 1
PNEUMONIA (Infections and infestations) | 1
ABDOMINAL PAIN DIARRHEA NAUSEA VOMITING (Gastrointestinal disorders) | 1
SEPSIS (Infections and infestations) | 1
ANEMIA (Blood and lymphatic system disorders) | 1
HYPERSENSITIVITY (Immune system disorders) | 1
NAUSEA VOMITING DYSPNEA (Gastrointestinal disorders) | 1
BILATERAL PULMONARY EMBOLISM (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Plitidepsin (N=24)
ANEMIA (Blood and lymphatic system disorders) | 7
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 3
CONSTIPATION (Gastrointestinal disorders) | 4
DIARRHEA (Gastrointestinal disorders) | 10
NAUSEA (Gastrointestinal disorders) | 19
VOMITING (Gastrointestinal disorders) | 7
EDEMA LIMBS (General disorders) | 6
FATIGUE (General disorders) | 22
FEVER (General disorders) | 5
INFUSION RELATED REACTION (General disorders) | 2
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER (General disorders) | 2
LUNG INFECTION (Infections and infestations) | 2
FRACTURE (Injury, poisoning and procedural complications) | 2
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2
ALKALINE PHOSPHATASE INCREASED (Investigations) | 2
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2
CARDIAC TROPONINE T INCREASED (Investigations) | 3
CPK INCREASED (Investigations) | 2
GGT INCREASED (Investigations) | 3
WEIGHT LOSS (Investigations) | 4
INVESTIGATIONS OTHER (Investigations) | 2
ANOREXIA (Metabolism and nutrition disorders) | 13
DEHYDRATATION (Metabolism and nutrition disorders) | 2
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 3
HYPOCALCEMIA (Metabolism and nutrition disorders) | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2
MYALGIA (Musculoskeletal and connective tissue disorders) | 5
HEADACHE (Nervous system disorders) | 3
NERVOUS SYSTEM DISORDERS OTHER (Nervous system disorders) | 2
INSOMNIA (Psychiatric disorders) | 2
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 5
RESPIRATORY THORACIC AND MEDIASTINAL DISORDERS OTHER (Respiratory, thoracic and mediastinal disorders) | 2
THROMBOEMBOLIC EVENT (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less